CLINICAL TRIAL: NCT02506049
Title: Fetoscopic Directed Laser Photocoagulation of Communicating Placental Vessels in Twin to Twin Transfusion Syndrome
Brief Title: Laser Photocoagulation in Twin to Twin Transfusion Syndrome
Acronym: TTTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee (Other)
Collaborators: Regional Medical Center, Regional One Health (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-00755-HUD
Record Dates: First submitted 2015-07-06; First posted 2015-07-22 (Estimated); Last update posted 2020-11-13 (Actual); Status verified 2019-01

CONDITIONS: Twin to Twin Transfusion Syndrome
MeSH Terms: conditions — Fetofetal Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- S-LPC:Selective Laser Photocoagulation (Other): S-LPC seals connecting vessels, normalizes flow between twins
  Interventions: Device: S-LPC:Selective Laser Photocoagulation

INTERVENTIONS:
Device: S-LPC:Selective Laser Photocoagulation — Under anesthesia (epidural, general anesthesia with intubation, or intravenous sedation with infiltration of a local anesthetic), one treatment with the use of fetoscopy instrument sets for Selective Laser Photocoagulation (S-PLC) to seal the connecting blood vessels, help to normalize blood flow between twins.

SUMMARY:
Humanitarian use device (HUD): Use of the fetoscopy instrument sets for selective laser photocoagulation in the treatment of Twin to Twin Transfusion Syndrome (TTTS).

DETAILED DESCRIPTION:
Patients initially will be identified by ultrasound examination by their primary provider. Consultation and subsequent ultrasound confirmation will be undertaken by our group. Patients meeting the inclusion criteria will undergo extensive verbal counseling regarding the clinical findings, prognosis, and management options. Those electing to proceed will sign written informed consent documents.

More specifically, after initial referral to our center for TTTS management, patients will undergo targeted ultrasound to confirm the diagnosis. If confirmed, patients will undergo extensive counseling regarding various management options. Those patients electing to proceed with selective laser photocoagulation (S-LPC) will undergo the informed consent process. The S-LPC will be performed in the Labor and Delivery (L&D), Operating Room (OR) at the Regional Medical Center, Regional One Health (RMC,ROH). In the majority of cases, maternal anesthesia will be an epidural. In those cases where the patient is unable to lay supine due to an enlarged uterus (resulting in maternal hypotension or respiratory insufficiency, or maternal anxiety), general anesthesia with intubation will be administered. In rare cases, intravenous sedation with infiltration of a local anesthetic into the skin, deep muscle, and fascia will be used. Following the administration of maternal anesthesia, ultrasound will be performed to assess fetal position, placentation, and select a site for insertion of the operative instruments. A small skin incision will be made following administration of local anesthetic to allow percutaneous access to the recipient gestational sac. An 18 gauge needle will be inserted through the maternal abdomen and uterus into the gestational sac. Once secured in place, the stylet will be removed and a J guide wire will be inserted through the needle. The needle will be removed and a 10-12 Fr (3-3.4 mm) trocar and cannula will be inserted into the sac over the guide wire. The trocar and guide wire will be removed and the fetoscopy instruments will be introduced through the cannula. The procedure is performed under continuous ultrasound guidance. After introduction of the fetoscope and operating sheath, the placenta is inspected by direct visualization for communicating vessels between the recipient and donor twin. A 400-600 micron laser fiber is introduced into the gestational sac via an instrument channel in the operating sheath. The fiber is directed to the communicating vessels, which are then ablated with thermal energy. An average of 7-15 sites will be ablated. At the completion of the procedure the amniotic fluid volume in the recipient sac will be reduced to a normal volume. Follow-up visits to track maternal and fetal progress after the procedure will be scheduled with our group.

ELIGIBILITY:
Inclusion Criteria:

* The device will be used in multifetal pregnancies affected with twin-to-twin transfusion syndrome (TTTS) at less than 27 weeks of gestation

Exclusion Criteria:

* All other pregnancies not meeting inclusion criteria

Ages: 16 Weeks to 27 Weeks | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2010-04; Primary Completion 2020-08-15 (Actual); Study Completion 2020-10-28 (Actual)

PRIMARY OUTCOMES:
Laser ablation of placental anastomoses for treatment of severe TTTS and establishment of normalized blood flow between the fetal twins. | The device will be used in multifetal pregnancies affected with twin-to-twin transfusion syndrome (TTTS) at less than 27 weeks of gestation;procedure will last approx 1 hour
  Once a diagnosis of TTTS has been made, the Fetoscopy Instrument Sets are intended to be used for selective laser photocoagulation (S-LPC) to treat the condition in fetuses whose gestational age is between 16 and 26 weeks. The set consists of a fetoscope, which is essentially an optical device used to view a fetus within the uterus, and sheaths that are used to pass other surgical instruments and/or fluid through the entry site, which is a tiny incision in the mother's abdomen. The instruments are inserted using ultrasound guidance and, once the shared blood vessels on the placenta are identified using the fetoscope, a laser can be passed through the sheath. The laser is used to photocoagulate the shared vessels. This helps to normalize the flow of blood between the twins. After all target vessels are identified and treated with S-LPC, the laser, fetoscope, and sheath are removed.

CONTACTS AND LOCATIONS:
Overall Officials: Giancarlo Mari, M.D., MBA, Principal Investigator — Prof. & Chair, UTHSC; Dir.,TN Inst. of Feto-Maternal & Infant Health; Dir., High-Risk Obstetrics Ctr of Excell., Regional Medical Ctr
Locations (2):
- United States (2):
  - Regional One Health, Regional Medical Center, Rout Center for Women and Children, Memphis, Tennessee
  - University of Tennessee Health Science Center, OB-GYN, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No